CLINICAL TRIAL: NCT05673317
Title: A Technological Approach to Improved Breastfeeding Rates and Self-Efficacy: A Randomized Controlled Clinical Trial
Brief Title: A Technological Approach to Improved Breastfeeding Rates and Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1505563
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Breastfeeding Self-Efficacy; Technology
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Control group received usual breastfeeding care (counseling by provider, access to lactation consultant, etc). Interventional received usual care plus the breastfeeding application introduced at the time of delivery or within 1 week postpartum.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participant cannot be blinded as they will be using the application.
  The investigator cannot be blinded as they have to provide the application to the patient, teach them how to use it, and perform their surveys about the application use.
  The outcomes assessor and care provider will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment Arm (Experimental): The participant will receive usual breastfeeding care such as counseling by her physician, access to lactation consults, nursing assistance in the hospital, access to our online resources. The participant will also receive the breastfeeding application at admission to labor and delivery or in the immediate postpartum period. The participant will be taught how to use the application, and will have access to the study to continue use throughout the duration of follow-up.
  Interventions: Other: "Breastfeeding at AU" Smartphone Application
- Control Arm (No Intervention): The participant will receive usual breastfeeding care such as counseling by her physician, access to lactation consults, nursing assistance in the hospital, access to our online resources.

INTERVENTIONS:
Other: "Breastfeeding at AU" Smartphone Application — This is a free Apple-Based Smartphone Application the participant can download. In the application, there is information and tips for breastfeeding success and continuation, as well as information on additional resources both online and in the community as a whole.
  Arms: Experiment Arm

SUMMARY:
To provide patients with easily accessible information in the form of a smartphone application regarding medically appropriate information about breastfeeding and to assess the impact this information has on women's breastfeeding rates and perception of self-efficacy (primary outcome).

DETAILED DESCRIPTION:
The benefits of breastfeeding for both mother and neonate have been well documented and extensively researched. Breastfeeding rates remain suboptimal despite known advantages including reduced lifetime risk of maternal ovarian cancer, more rapid return to pre-gestational weight, improvement in maternal/neonatal bonding, reduction in neonatal allergic/immunologic conditions. Both non-modifiable and modifiable factors affecting a mother's decision regarding breastfeeding have been identified. Modifiable factors include breastfeeding knowledge, self-efficacy, and confidence. Breastfeeding self-efficacy has been positively correlated with breastfeeding duration. There is a lack of local data on breastfeeding rates, duration, and self-efficacy in the Augusta University women's health population as well as a lack of documented improvement of these factors following educational programs. Our study aims to create a program that is easily accessible and available to our patient population in the form of a free application available on Apple devices capable of accessing the internet (e.g., i-phone, i-pad, etc.). This study will be a randomized controlled pilot study. The intervention group will have access to the application while the control group will not. Our hypothesis is that the application will improve breastfeeding rates, duration, and self-efficacy if offered to at the time of delivery or within the first week postpartum. This will be assessed by comparing initial self-efficacy survey results (within 1 week postpartum) with survey results at 4 to 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Patients intending to breastfeed receiving prenatal care at Augusta University.
* No documented anatomic differences in mother's chest anatomy.
* Access to the internet via an Apple® device (such as i-phone or i-pad).
* Delivery at Augusta University Medical Center

Exclusion Criteria:

* Significant maternal intrapartum or postpartum complications (i.e., postpartum hemorrhage > 2000 mL, uterine inversion, retained products, ICU admission, postpartum psychosis).
* Infants admitted to neonatal intensive care unit >48 hours
* Pre-term deliveries prior to 37 weeks gestation
* Infants with cleft palate, or other palate/facial defects
* Patients without email access or internet access
* Patients without an Apple® device (i-phone, i-pad)
* Non-English speaker
* Patients unable to breastfeed secondary to contraindicated communicable disease (i.e.

HIV)

* Patients unable to breastfeed secondary to contraindicated medications
* Patients of infants up for adoption

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be a genotypic female who gave birth with intention to breastfeed their infant to participate in this study.
Enrollment: 40 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Score | 6 weeks
  The breastfeeding self-efficacy short form is a validated, standardized form to assess participants' sense of breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Breastfeeding rate | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: 5 years after the study
Access Criteria: Email czahlermiller@augusta.edu